CLINICAL TRIAL: NCT04791215
Title: An Observational Study of Circulating Tumor DNA Genetic Alterations in Non-small Cell Lung Cancer Patients Treated With Pembrolizumab
Brief Title: Circulating Tumor DNA Alterations in Non-small Cell Lung Cancer Patients Treated With Pembrolizumab
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAS7953
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Cancer; Immune system; Lung Cancer; Pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and residual tissue from surgery or tumor biopsy will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Sample Collection: Prospective sample collection from participants treated with pembrolizumab monotherapy at Columbia University Irving Medical Center under standard of care treatment. Prospective cohort subjects must consent to provide available archived tumor and blood for whole exome sequencing (WES) (matched tumor and normal) for creation of plasma ctDNA panels. The tumor sample must be from a site that was not previously irradiated or has progressed after radiation.
  Interventions: Other: Observational
- Retrospective Sample Collection: Retrospective sample collection from participants that consent to provide genetic data from previous whole exome sequencing (WES) in the form of files for creation of plasma ctDNA panels.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — All patients will be treated with standard of care pembrolizumab. After obtaining written informed consent, NSCLC participants will have serial blood collection. The blood collection (26 ml) should coincide with routine clinical blood draw to minimize participant discomfort if possible. No additional procedures will be performed other than phlebotomy. If additional biopsies or tumor resection are performed as part of routine standard of care throughout the course of the study, an additional 26 ml blood collection may be drawn for the study. Participants will remain on the study for as long as they are being followed or treated at Columbia University Irving Medical Center. Participants can withdraw from the study at any time.

SUMMARY:
The purpose of this study is to learn how to use blood tests to better predict how patients with non-small cell lung cancer, who are taking pembrolizumab for cancer treatment, will respond to treatment with pembrolizumab, and to understand how the immune system and cancer interact.

Tests will be performed on tumor tissue and blood samples, and imaging assessments will be reviewed in order to monitor how well each patient responds to treatment. This is an observational study, so participants will not receive cancer treatment, other than the treatment received as standard of care.

DETAILED DESCRIPTION:
The primary and secondary endpoints of this study are to determine the kinetics of Circulating tumor DNA (ctDNA) as defined by a set of patient-specific tumor mutations. The analysis will be undertaken using the Signatera Assay from Natera. Circulating tumor DNA in plasma samples obtained over the course of pembrolizumab treatment will be assessed by high-intensity, next-generation genetic sequencing to identify genomic alterations in genes. The assay will target 16 defined patient specific mutations. Data acquired will be analyzed to characterize the association between these genetic elements, clinical response, and durability of responses. There will be prospective and retrospective groups for the study. Samples will be collected from patients in the prospective cohort who have been treated with pembrolizumab monotherapy at Columbia University Irving Medical Center under standard of care treatment. Subjects in the retrospective cohort will provide genetic data.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of NSCLC with a protein that acts as a kind of "brake" to keep the body's immune responses under control called Programmed Death Ligand-1 (PD-L1) Tumor Proportion Score (TPS) ≥ 1% and no known alterations in driver genes epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or receptor tyrosine kinase (ROS1).
2. Retrospective cohort: subjects must consent to provide genetic data from previous whole exome sequencing (WES) in the form of FASTQ/BAM files (files that represent aligned genetic sequences) for creation of plasma ctDNA panels.
3. Prospective cohort: Subjects must consent to provide available archived tumor and blood for WES (matched tumor and normal) for creation of plasma ctDNA panels. The tumor sample must be from a site that was not previously irradiated or has progressed after radiation.
4. Ability to understand and the willingness to sign a written informed consent document.
5. Willing to comply with clinical trial instructions and requirements.
6. Both men and women of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

1. Age <18 years
2. Known history of autoimmune disease or other medical conditions that would preclude safe treatment with pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male and females with a diagnosis of NSCLC with a protein that acts as a kind of "brake" to keep the body's immune responses under control PD-L1 TPS ≥1% and no known alterations in driver genes epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or Proto-oncogene tyrosine-protein kinase (ROS1).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Radiologic response to immune checkpoint blockade (ICB) by clonal dynamics of serial ctDNA in 1st line NSCLC patients receiving pembrolizumab monotherapy. | 5 years
  Radiologic response to immune checkpoint blockade (ICB) by clonal dynamics of serial ctDNA in 1st line NSCLC participants receiving pembrolizumab monotherapy. Imaging studies will be performed per RECIST 1.1. Radiologic response measured as the average time between randomization and detection of overt progression or response by ctDNA compared to RECIST 1.1.

SECONDARY OUTCOMES:
To characterize kinetic profiles of tumor mutations and see if they are predictive of overall survival (OS) and progression-free survival (PFS). | 5 years
  To characterize kinetic profiles of defined tumor mutations in tumor fraction ctDNA and evaluate whether they are predictive of overall survival (OS) and progression-free survival (PFS). A blood-based ctDNA assay offers the advantage of a read-out of these temporal changes, with the prospect of kinetic assessment of tumor fraction ctDNA being predictive for early response or progression to immunotherapy. The ability to assess temporal changes in tumor genetics will give insight into tumor clonal evolution and immune editing of specific neoantigens, which may enable leveraging of these insights for future diagnostic and therapeutic improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Henick, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided